CLINICAL TRIAL: NCT00007735
Title: CSP #475 - Persian Gulf - Antibiotic Treatment Trial of Gulf War Veterans' Illnesses
Brief Title: Antibiotic Treatment of Gulf War Veterans' Illnesses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Pfizer (Industry); United States Department of Defense (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 475
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2007-02

CONDITIONS: Persian Gulf Syndrome; Mycoplasma Infections
Keywords: antibiotic treatment; mycoplasma species; Gulf War Veterans' Illnesses (GWI); mycoplasma positive; Gulf War Syndrome
MeSH Terms: conditions — Persian Gulf Syndrome; Mycoplasma Infections | interventions — Doxycycline

INTERVENTIONS:
Drug: Doxycycline (200mg/day) or Placebo

SUMMARY:
In 1990 and 1991, the U.S. deployed approximately 700,000 troops to the Persian Gulf to liberate Kuwait from Iraqi occupation. While there were few casualties associated with the Gulf War, many individuals returned from this conflict with unexplained symptoms and illnesses. This constellation of symptoms has been termed Gulf War Veterans' Illnesses (GWI). Although several explanations have been offered as to the cause of GWI, none of the putative etiologic agents or conditions is currently supported by sufficient evidence. One explanation that has received fairly widespread attention is systemic Mycoplasma fermentans infection. It is the purpose of this study to determine if antibiotic treatment directed against Mycoplasma species (i.e. doxycycline) will improve functioning and symptoms in deployed Gulf War veterans with GWI.

DETAILED DESCRIPTION:
Primary Hypothesis: The primary hypothesis of this study is that antibiotic treatment directed against Mycoplasmaspecies will improve functional status of patients with Gulf War Veterans' Illnesses (GWI) who are tested as mycoplasma positive at baseline. Specifically, the primary objective of the study is to determine whether a 12 month course of doxycycline treatment in deployed Gulf War veterans presenting with symptoms of GWI and testing as mycoplasma positive improves functional status compared to placebo.

Secondary Hypotheses: Secondary objectives of this study are (1) to determine whether doxycycline treatment reduces symptoms of GWI including pain, fatigue and neurocognitive concerns, (2) to determine whether doxycycline treatment converts mycoplasma positive patients to mycoplasma negative status, and (3) to determine if the benefits of 12 months doxycycline treatment persist after termination of treatment.

Intervention: Patients are randomized to either doxycycline (200mg/day) or placebo which they are instructed to take in the morning.

Primary Outcomes: The primary outcome measure is improvement in the Physical Component Scale (PCS) of the SF-36V at follow-up relative to baseline. The primary end point will be the proportion of patients with more than a seven unit increase in the PCS at 12 months. Important secondary outcome measures are a pain scale (McGill Pain Questionnaire), a fatigue scale (Multidimensional Fatigue Inventory), a neurocognitive symptoms scale (Cognitive Failures Questionnaire), and a GWI Symptom Checklist developed specifically for this study.

Study Abstract: In 1990 and 1991, the U.S. deployed approximately 700,000 troops to the Persian Gulf to liberate Kuwait from Iraqi occupation. While there were few casualties associated with the Gulf War, many individuals returned from this conflict with unexplained symptoms and illnesses. This constellation of symptoms has been termed Gulf War Veterans' Illnesses (GWI). Although several explanations have been offered as to the cause of GWI, none of the putative etiologic agents or conditions is currently supported by sufficient evidence. One explanation that has received fairly widespread attention is systemic Mycoplasma fermentans infection. It is the purpose of this study to determine if antibiotic treatment directed against Mycoplasma species (i.e. doxycycline) will improve functioning and symptoms in deployed Gulf War veterans with GWI.

The study is a 30 month, prospective, randomized, double-blind clinical trial. All veterans deployed to the Gulf War between August, 1990 and August, 1991 will be eligible. Patients will be considered to have GWI if they have at least two of three symptoms (fatigue, musculoskeletal pain, neurocognitive dysfunction) that began after August, 1990 and that have lasted more than six months up to the present. Four hundred and fifty of these GWI patients from 28 medical centers who test positive for Mycoplasma fermentans, Mycoplasma gentalium and/or Mycoplasma pneumoniae at baseline and have no exclusion criteria will be entered into the study over a one year recruitment period. These mycoplasma positive species patients will be randomized to one of two treatment groups: (1) patients treated with doxycycline for 12 months and (2) patients given placebo for 12 months. Each patient will receive study medication for 12 months and will be followed for an additional six months after the termination of medications. Patients will be seen monthly during the medication phase and at 18 months. Major evaluations will be completed at baseline and at 3, 6, 9, 12 and 18 months. Patients assigned to doxycycline will receive 200mg/day, which they will be instructed to take in the morning.

MAIN MANUSCRIPT - Submitted to New England Journal of Medicine on February 22, 2002. On May 10, 2002, New Englad Journal of Medicine rejected the manuscript. Manuscript was submitted to LANCET on June 17, 2002 and rejected on July 29, 2002. Manuscript was submitted to JAMA on August 30, 2002 and rejected on September 6, 2002. Manuscript has been resubmitted to JAMA on March 24, 2003.

ELIGIBILITY:
All veterans deployed to the Gulf War between August, 1990 and August, 1991 having at least two of the following symptoms: Fatigue, musculoskeletal pain or neurocognitive dysfunction. Mycoplasma positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 1999-01; Study Completion 2001-10

CONTACTS AND LOCATIONS:
Locations (27):
- United States (26):
  - Vamc - Birmingham, Al, Birmingham, Alabama
  - Naval Health Research Center Merchant Illness Divi, San Diego, California
  - Uniformed Services University Department of Psychi, Washington D.C., District of Columbia
  - Vamc - Augusta, Ga, Augusta, Georgia
  - Vamc - Hines,Il, Hines, Illinois
  - Vamc - New Orleans, La, New Orleans, Louisiana
  - Vamc - Boston, Ma, Boston, Massachusetts
  - Vamc - Omaha, NE, Omaha, Nebraska
  - Vamc - Manchester,Nh, Manchester, New Hampshire
  - Vamc - East Orange, Nj, East Orange, New Jersey
  - Vamc - Albuquerque, Nm, Albuquerque, New Mexico
  - Vamc - Albany, Ny, Albany, New York
  - Vamc - Brooklyn, Ny, Brooklyn, New York
  - Vamc - Bronx,Ny, The Bronx, New York
  - Vamc - Durham, Nc, Durham, North Carolina
  - Vamc - Fargo, Nd, Fargo, North Dakota
  - Vamc - Dayton, Oh, Kettering, Ohio
  - Vamc - Oklahoma City, Ok, Oklahoma City, Oklahoma
  - Vamc - Philadelphia, Pa, Philadelphia, Pennsylvania
  - Vamc - Providence, Ri, Providence, Rhode Island
  - Vamc - Charleston, Sc, Charleston, South Carolina
  - Vamc - Nashville, Tn, Nashville, Tennessee
  - Vamc - Houston, Tx, Houston, Texas
  - Vamc - White River Junction, White River Junction, Vermont
  - Vamc - Richmond, Va, Richmond, Virginia
  - Vamc - Milwaukee, Wi, Milwaukee, Wisconsin
- Vamc - San Juan, Pr, San Juan, Puerto Rico